CLINICAL TRIAL: NCT04290689
Title: Can Gait Analysis and Imaging Methods Detect Change in the Calf Musculature in Children With Cerebral Palsy? Comparison Study of Toe Walking Patients Following Serial Casting, Botulinum Toxin-A and Typically Developing Controls.
Brief Title: Can Gait Analysis and Ultrasound Detect a Change in Calf Musculature in Children With Cerebral Palsy?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1 777
Record Dates: First submitted 2019-10-29; First posted 2020-03-02 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; b-mode ultrasound; gait analysis; EMG; elastography; musculoskeletal modelling
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Botulinum Toxin-A injection treatment: Toe walking Cerebral Palsy subject who are subject to Botulinum toxin-A injection treatment. The dosage will be determined by the Orthopaedic Consultant
  Interventions: Drug: Botulinum Toxin-A injection
- Serial casting stretching treatment: Toe walking Cerebral Palsy subject who are subject to serial casting stretching treatment.
  Interventions: Procedure: Serial casting stretching

INTERVENTIONS:
Drug: Botulinum Toxin-A injection — Botulinum Toxin-A injection to be administered by the surgeon to the subject's calf muscle as per normal clinical protocol to help improve muscle tone.
  Other Names: "Botox"
  Groups: Botulinum Toxin-A injection treatment
Procedure: Serial casting stretching — Stretching cast intervention to be carried out in clinic as per normal clinical protocol.
  Other Names: serial cast
  Groups: Serial casting stretching treatment

SUMMARY:
ORLAU is a clinical department of the Robert Jones and Agnes Hunt Orthopaedic Hospital. We treat patients with a wide range of movement disorders affecting their walking or arm function. One of the most common gait issues we see is toe-walking, this is most prevalent in those patients with cerebral palsy (CP). Toe-walking in CP children arises mostly from problems in the calf muscle, we currently use gait analysis to help guide treatment management plans. Two standard interventions for such cases are serial casting and Botulinum Toxin-A injections. Using gait analysis we will be able to see changes to the gait pattern before and after the interventions, however, we want to obtain a whole clinical picture, using B-mode ultrasound, elastography and electromyography (EMG) we will be able to achieve this. These measurements will provide us with information about the muscle architecture and properties including activation. This will help us to determine the effects of the interventions. Elastography is a fairly new clinical technique that uses shear waves generated by the ultrasound probe to map the stiffness of a muscle. Stiffness of muscle is a good indication of myopathies. The additional examinations we want to carry out are all non-invasive, they will be carried out in two sessions, one before the intervention and one after. We will compare the data we collect from the children with CP to our normal database with ORLAU has ethical approval for. The final stage of this study will be to use the muscle parameters obtained by ultrasound to set parameters in a computer musculoskeletal model.

DETAILED DESCRIPTION:
The aim of this study is to investigate the impact on gait and morphology of the calf muscle in children with Cerebral Palsy with equinus gait pattern following serial casting and Botulinum toxin (Btx) interventions.

Toe walking is a common feature of a number of orthopaedic and neurological problems (e.g. cerebral palsy, idiopathic toe walking and stroke). Patients who toe walk often develop contractures in their calf muscles and in the longer term may suffer from foot or calf pain and foot deformities. Toe walking also causes difficulties with balance and leads to secondary compensations and deformities. The causes of toe walking are not always clear for individual patients. Current interventions target the perceived causes (e.g. surgery, stretching or orthotics for contracture or botulinum toxin injections for excessive activity) but the relationship between toe walking and the impairment in muscle morphology and control is not fully understood. Clinical movement analysis is used to quantify joint motion and loading during gait. This is done according to established local departmental protocol and is part of routine clinical practice. This is done using the Video Based Motion Analysis System Ltd (VICON), which is a 3D movement analysis modality which makes use of small, spherical reflective markers, between 5mm and 25mm in diameter that are attached to the skin over key anatomical landmarks (located during the clinical examination). Special infrared cameras are used to track the movements of reflective markers in three dimensions. This is combined with AMTI force plates; which together give the kinematics and kinetics of the subject. Electromyography (EMG) of the Triceps Surae and Tibialis Anterior enables observation of muscle activity in conjunction with the gait cycle during different movements. After obtaining participant consent and ensuring that the participant fully understands the scope of the tasks, the session is undertaken. In brief, using local ORLAU department protocol, a clinician places reflective markers on the subject and anthropometric measurements are taken. After the subject is prepared, they are asked to walk along a 10-metre walkway at a self selected speed and a minimum of 6 trials are collected with adequate strikes with each foot landing on the force plate to obtain desired kinematic and kinetic data. EMG recordings are performed simultaneously on the Medial & Lateral Gastrocnemius, Soleus, and Tibialis Anterior to record muscle activity during the movement.

To obtain information about the morphology, the modality of B-mode ultrasound evaluated the muscle morphology and obtains key information such as muscle fibre length, fibre orientation, pennation angle, cross sectional area, and muscle thickness. After obtaining consent and ensuring that the participant understands fully the scope of the session, they are asked to lie prone on the plinth with lower legs exposed so that the assessor has access to the calf muscles. The assessor then uses the b-mode ultrasound protocol to obtain the key parameters of the calf muscle. Muscle lengths are measured using a Vernier caliper.

In addition, the imaging modality elastography is used. This uses mechanical force, from manual pressure or through a shear wave impulse generated within the ultrasound probe, to detect the change in deformation of the examined tissue and therefore to determine the stiffness. The stiffness of soft tissues can be an indication of pathology. Elastography uses harmless ultrasound waves and allows for the visualisation of strain across a tissue, by superimposing the colour coded elasticity map onto a conventional B-mode image. The colours represent the stiffness of the tissue ranging from red to green to blue, with the exact scale varying between vendors. Shear wave elastography has the added advantage of being able to provide velocity measurements within a defined region of interest, thus quantifying tissue stiffness.

Prior to beginning the session, consent from the subject is obtained and the scope of the session is explained. After consent from the participant, the subject is asked to lie prone on the plinth with their lower legs exposed. The consultant radiologist undertakes elastography measures on the calf muscles (medial, lateral gastrocnemius, soleus) in longitudinal and transverse planes according to the protocol. These are then saved after the key information is obtained and analysed after the session.

Computer modelling can estimate muscle forces during gait, and it is used to study a wide range of conditions such as spastic paresis and crouch gait. Ultrasound can provide information about muscle parameters such as volume, length, anatomical cross-sectional area and pennation angle. This information can be used to adjust the parameters of the musculoskeletal model to fit the characteristics of each patient. The musculoskeletal model can then estimate personalised muscle forces and help understand the individual impairments which lead to toe walking. Future prospects Clinical- The computer models will assist with the precise identification of impairments (eg muscle atrophy, contracture and spasticity) and hence allow more objective specification and targeting of interventions. Combining the data collected from B mode ultrasound, elastography and gait analysis, the effects of clinical interventions in muscle properties can be observed. This can be applied to other interventions, including orthopaedic surgery and orthotic devices. Elastography can also be a vital tool in understanding the elastic muscle properties associated with myopathies and can help optimise and personalise care by selecting the most effective intervention based on an individual's baseline features.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with Cerebral Palsy and have a planned intervention of serial casting or botulinum toxin calf injection or serial casting and botulinum toxin injection.
* Participants must be able to walk 10 metres barefoot.
* Participants must be between the ages of 4 and 16.
* Participants must have a gait pattern showing persistent toe walking or premature heel rise.
* Participants should be able to comply with requests to walk in the gait laboratory.

Exclusion Criteria:

* Participants who have had Botulinum toxin-A calf injections or previous serial casting within the last 6 months.
* Participants should not have fixed foot equinus.
* Participants must not have any learning difficulties which would prevent compliance with the standard protocols.
* Participants must not have had any previous surgical interventions of the lower limbs within one year of taking of taking part.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Potential participants will be screened by the research team at weekly review meeting (involving the Medical Director and orthopaedic consultants). Participants will be identified in the Childrens outpatient's clinics at Trust Hospital (RJAH).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-03-14 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Are there gait (kinetic) differences pre and post intervention in toe walking cerebral palsy subjects? | up to12 weeks
  Kinetics (joint forces) will be measured (using gait analysis modality) pre and post intervention in toe walking cerebral palsy subjects. The intervention will be determined by the consultant Orthopedic Surgeon in clinic.Units of measure:measured in Nm/kg
Are there gait (kinematic) differences pre and post intervention in toe walking cerebral palsy subjects? | up to 12 weeks
  Kinematics (joint angles) will be measured (using gait analysis modality) pre and post intervention in toe walking cerebral palsy subjects. The intervention will be determined by the consultant Orthopedic Surgeon in clinic.Units of measure: measured in degrees (angle).
Triceps Surae muscle activation during the gait cycle (Electromyography) | up to12 weeks
  Electromyography (EMG) measurement - is the muscle activated or deactivated pre and post intervention in toe walking cerebral palsy subjects? Measured in uV
Are there morphological differences in the calf muscle pre and post serial casting/botulinum toxin-A intervention in toe walking cerebral palsy subjects? | up to 12 weeks
  B-mode ultrasound modality will be used pre and post intervention to measure muscle morphology parameter - muscle thickness. Measured in millimeter
Are there morphological differences in the calf muscle pre and post serial casting/botulinum toxin-A intervention in toe walking cerebral palsy subjects? | up to 12 weeks
  B-mode ultrasound modality will be used pre and post intervention to measure muscle morphology parameter - muscle fibre length; measured in millimeter
Are there morphological differences in the calf muscle pre and post serial casting/botulinum toxin-A intervention in toe walking cerebral palsy subjects? | up to 12 weeks
  B-mode ultrasound modality will be used pre and post intervention to measure muscle morphology parameter - muscle length; measured in millimeter
Are there morphological differences in the calf muscle pre and post serial casting/botulinum toxin-A intervention in toe walking cerebral palsy subjects? | up to 12 weeks
  B-mode ultrasound modality will be used pre and post intervention to measure muscle morphology parameter - pennation angle; measured in degrees.
Are there morphological differences in the calf muscle pre and post serial casting/botulinum toxin-A intervention in toe walking cerebral palsy subjects? | up to 12 weeks
  B-mode ultrasound modality will be used pre and post intervention to measure muscle morphology parameter - Cross sectional area; measured in cm^2
Difference in the muscle stiffness values (using elastography) in the calf muscle pre and post intervention. | up to 12 weeks
  To determine, using elastography modality, if there is a difference in muscle stiffness values pre and post intervention for toe walking cerebral palsy children. Units of measure: m/s velocity

OTHER OUTCOMES:
Are there gait (kinetic and kinematic) differences pre and post intervention in toe walking cerebral palsy subjects? | up to 12 weeks
  The temporospatial parameter during the gait analysis will be measured pre and post intervention: walking speed; units of measure:m/s
Are there gait (kinetic and kinematic) differences pre and post intervention in toe walking cerebral palsy subjects? | up to 12 weeks
  The temporospatial parameter during the gait analysis will be measured pre and post intervention: cadence; units of measure: steps/min
Are there gait (kinetic and kinematic) differences pre and post intervention in toe walking cerebral palsy subjects? | up to 12 weeks
  The temporospatial parameter during the gait analysis will be measured pre and post intervention: single/double support ; units of measure: single/double
Are there gait (kinetic and kinematic) differences pre and post intervention in toe walking cerebral palsy subjects? | up to 12 weeks
  The temporospatial parameter during the gait analysis will be measured pre and post intervention:step width; units of measure: meter

CONTACTS AND LOCATIONS:
Locations (1):
- ORLAU, RJAH Orthopaedic Hospital, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Study is still recruiting and collecting data. sharing will depend on the quality and quantity of data collected.

REFERENCES:
- [Background] Armand S, Decoulon G, Bonnefoy-Mazure A. Gait analysis in children with cerebral palsy. EFORT Open Rev. 2016 Dec 22;1(12):448-460. doi: 10.1302/2058-5241.1.000052. eCollection 2016 Dec. PMID 28698802
- [Background] Barber L, Barrett R, Lichtwark G. Passive muscle mechanical properties of the medial gastrocnemius in young adults with spastic cerebral palsy. J Biomech. 2011 Sep 2;44(13):2496-500. doi: 10.1016/j.jbiomech.2011.06.008. Epub 2011 Jul 16. PMID 21762920
- [Background] Blemker SS, Asakawa DS, Gold GE, Delp SL. Image-based musculoskeletal modeling: applications, advances, and future opportunities. J Magn Reson Imaging. 2007 Feb;25(2):441-51. doi: 10.1002/jmri.20805. PMID 17260405
- [Background] Stewart C, Shortland AP. The biomechanics of pathological gait - from muscle to movement. Acta Bioeng Biomech. 2010;12(3):3-12. PMID 21247058
- [Background] Kalsi G, Fry NR, Shortland AP. Gastrocnemius muscle-tendon interaction during walking in typically-developing adults and children, and in children with spastic cerebral palsy. J Biomech. 2016 Oct 3;49(14):3194-3199. doi: 10.1016/j.jbiomech.2016.07.038. Epub 2016 Aug 8. PMID 27545082